CLINICAL TRIAL: NCT06062147
Title: Prevention, Detection and Specialised Intervention in Pre-school : Impact of Teacher Training and the Introduction of Early Adjustments on the Developmental Trajectory of Children at Risk of Specific Language and Learning Disorders (SLLD).
Brief Title: Impact of Teacher Training and the Introduction of Early Adjustments on the Developmental Trajectory of Children at Risk of SLLD in Pre-school.
Acronym: PRISME-TSLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023/CHU/28; 2023-A01501-44 (Other: ID-RCB)
Record Dates: First submitted 2023-09-22; First posted 2023-10-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Language Disorders in Children; Learning; Developmental Disorder
Keywords: Professional development; Preventive approach; Neurological Development; Preschool education
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Pragmatic cluster controlled trial (quasi-experimental design)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- teacher training (Experimental): Teacher training and support for teachers in setting up specific arrangements.
  Interventions: Behavioral: Teacher training
- control class (No Intervention): Teacher will proceed in the usual way, referring to the procedures put in place by the national education system for identifying and referring children at risk

INTERVENTIONS:
Behavioral: Teacher training — Training for teachers in the intervention arm in the learning process, SLLD and early warning signs, with an identification grid. Observation of identified pupils and implementation of educational and environmental adjustments.
  Arms: teacher training

SUMMARY:
The high incidence of neurodevelopmental disorders, including specific language and learning disorders, and their profund impact on the schooling of the children concerned remains a major public health concern. Early identification and intervention are a valuable tool for improving these problems. The developmental trajectory of children could be improved by knowledge enhancement, identification and strategies to support the teachers through the involvement of health professionals in the classroom

DETAILED DESCRIPTION:
PRISME - TSLA is a clinical trial developing experiment project for the intervention arm involving teacher training, the implementation of identification grids, follow-up observations in classroom of identified pupils, and the development of special arrangments. For the control arm, the teachers work with standard procedures of the French national education policy.

ELIGIBILITY:
Inclusion Criteria:

Pupils :

* In a kindergarten school with at least 3 classes of primary school age children.
* At least 5 years old on 31/12/2023.
* Whose 2 parents have given their consent (the consent of a single parent if no contact is possible with the second parent despite repeated attempts)
* Have received age-appropriate explanations about the study and have not refused to take part.

Exclusion Criteria:

Pupils in :

* In a kindergarten school with fewer than 3 classes, making it impossible to randomise the school
* Under 5 years of age on 31 December of the current school year.
* Under guardianship

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Improvement in the developmental trajectory of pre-school children at risk of SLLD in the areas of language, learning and coordination | 8 months after inclusion
  BMTi (Modular Computerized Test Battery). pathologic area if score < or = -2, risk area if score [-1;-2[ middle area if score ]-1;1[ higher area if score > or = 1

SECONDARY OUTCOMES:
Improvement in teachers' knowledge and sense of competence | 8 months after inclusion
  knowledge quiz

CONTACTS AND LOCATIONS:
Overall Officials: Magali CARBONNNIER, MD, Principal Investigator — Fondation Père FAVRON
Locations (1):
- CHU de La Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No